CLINICAL TRIAL: NCT06968130
Title: Evaluation of the Effects of Virtual Reality Glasses and Respiratory Exercises on Symptoms and Quality of Life Among Patients Receiving Hemodialysis Treatment
Brief Title: Effects of Virtual Reality and Breathing Exercises on Hemodialysis Patients' Symptoms and Quality of Life
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ecehan Bulut, PhD student, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TÜTF-BAEK-2021/01
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Kidney Diseases
Keywords: Hemodialysis; quality of life; general assessment of symptoms; virtual reality; breathing exercise
MeSH Terms: conditions — Kidney Diseases | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Sham Comparator): Patients will receive routine hemodialysis without any additional intervention. The same scales will be administered at baseline and during two follow-ups one week apart.
  Interventions: Behavioral: routine hemodialysis
- Breathing Exercise Group (Active Comparator): Patients will perform deep breathing exercises guided by the researcher: 1 minute normal breathing, 3 minutes chest breathing, 3 minutes diaphragmatic breathing, 2 minutes pursed-lip breathing, and 1 minute normal breathing. Exercises will be conducted for 10 minutes before and after hemodialysis, repeated in two follow-up sessions one week apart, with post-session scale completion.
  Interventions: Behavioral: routine hemodialysis; Behavioral: Breathing Exercise
- Virtual Reality Group (Active Comparator): After completing the initial scales, patients will watch a 20-minute nature simulation via virtual reality glasses before and after hemodialysis. This will be repeated in two follow-up sessions one week apart, followed by scale administration.
  Interventions: Behavioral: routine hemodialysis; Device: Virtual Reality

INTERVENTIONS:
Behavioral: routine hemodialysis — Patients will receive routine hemodialysis without any additional intervention. The same scales will be administered at baseline and during two follow-ups one week apart.
Behavioral: Breathing Exercise — Patients will perform deep breathing exercises guided by the researcher: 1 minute normal breathing, 3 minutes chest breathing, 3 minutes diaphragmatic breathing, 2 minutes pursed-lip breathing, and 1 minute normal breathing. Exercises will be conducted for 10 minutes before and after hemodialysis, repeated in two follow-up sessions one week apart, with post-session scale completion.
  Arms: Breathing Exercise Group
Device: Virtual Reality — After completing the initial scales, patients will watch a 20-minute nature simulation via virtual reality glasses before and after hemodialysis. This will be repeated in two follow-up sessions one week apart, followed by scale administration.
  Arms: Virtual Reality Group

SUMMARY:
Purpose: This study aims to examine the effects of virtual reality glasses and breathing exercises on symptoms and quality of life in patients receiving hemodialysis treatment.

Design: This randomized controlled cross-sectional study will be conducted in the hemodialysis units of 3 state and 2 private hospitals. Individuals over 18 years old, diagnosed with End-Stage Renal Disease (ESRD), on hemodialysis for at least 3 months, without communication barriers, and volunteering to participate will be included. A power analysis using G*Power (v3.1.7) determined a sample size of 53 individuals per group for 80% power at α=0.05. Data will be collected through a demographic questionnaire, Dialysis Symptom Index (DSI), and WHOQOL-Bref-TR, with permission obtained from scale developers.

Participants will be randomized into three groups:

Experiment 1 (Virtual Reality Group): After completing the initial scales, patients will watch a 20-minute nature simulation via virtual reality glasses before and after hemodialysis. This will be repeated in two follow-up sessions one week apart, followed by scale administration.

Experiment 2 (Breathing Exercise Group): Patients will perform deep breathing exercises guided by the researcher: 1 minute normal breathing, 3 minutes chest breathing, 3 minutes diaphragmatic breathing, 2 minutes pursed-lip breathing, and 1 minute normal breathing. Exercises will be conducted for 10 minutes before and after hemodialysis, repeated in two follow-up sessions one week apart, with post-session scale completion.

Control Group: Patients will receive routine hemodialysis without any additional intervention. The same scales will be administered at baseline and during two follow-ups one week apart.

Statistics: Data analysis will be performed using Statistical Package for the Social Sciences (SPSS) Software. Descriptive statistics (mean, standard deviation, median, frequency, ratio) will be used. The Shapiro-Wilk test and box plot graphics will assess normality. For comparisons: ANOVA, Kruskal-Wallis H test, Tukey's post-hoc test, Pearson's chi-square test, Fisher's exact chi-square test, Bonferroni test, and multiple regression model analyses.

Significance will be set at p<0.05.

DETAILED DESCRIPTION:
Purpose: This study was planned to examine the effects of virtual reality glasses and breathing exercise applications on symptoms and quality of life in patients receiving hemodialysis treatment.

Design: This randomized controlled cross-sectional study will be applied to individuals diagnosed with End-Stage Renal Disease (ESRD) who were treated in hemodialysis units of 3 state hospitals and 2 private hospitals. No randomized controlled study was found using scales on patients diagnosed with ESRD in the literature review. Power analysis was performed using the G*Power (v3.1.7) program to determine the sample size. It was decided that there should be 53 people in the groups for 80% power at α=0.05 level.

People over the age of 18, diagnosed with end-stage renal disease, on hemodialysis for the last 3 months, without communication barriers and volunteering to participate in the study will be included in the study according to the randomization table.

The data will be filled with a questionnaire form containing demographic data, the Dialysis Symptom Index (DSI) and the World Health Organization Quality of Life Scale Short Form Turkish Version (WHOQOL-Bref-TR). Necessary permissions have been obtained from the people who developed the scales.

Patients who meet the research criteria will be assigned to experiment 1 (virtual reality glasses), experiment 2 (breathing exercise) and control groups according to the randomization table. Then;

1. Experiment 1 Group 1st Application: After the patients who agree to participate in the study sign the informed consent form, the demographic characteristics of the patients, the DSI and WHOQOL-Bref-TR scales will be filled in by the researcher. The patients will watch a simulation consisting of forest and nature images with virtual reality glasses for a total of 20 minutes before and after hemodialysis.

   In the 2nd and 3rd Applications, the patients will watch the same simulation at one-week intervals and then the DSI and WHOQOL-Bref-TR will be filled in.
2. Experiment 2 Group:

The researcher will demonstrate deep breathing exercises in a specific order and have the individuals apply the exercises one-on-one.

Procedure steps:

1. Normal breathing for 1 minute,
2. Chest breathing 20-24 times (approximately 3 minutes),
3. Diaphragmatic breathing (inhale through the nose and exhale through the nose) 20-24 times (approximately 3 minutes),
4. Pursed lip breathing 16-20 times (approximately 2 minutes) (inhale through the nose and exhale through the mouth),
5. Normal breathing for 1 minute

1. Application: After the patients who agree to participate in the study sign the informed consent form, the demographic characteristics of the patients, DSI and WHOQOL-Bref-TR scales will be filled out by the researcher. The patients will be applied a total of 10 minutes of exercises before and after hemodialysis.

In the 2nd and 3rd applications, the patients will be subjected to the same breathing exercise one week apart and then the DSI and WHOQOL-Bref-TR will be filled in.

3rd Control Group:

1. st Application: After the informed consent form is signed by the patients who agree to participate in the study, the demographic characteristics of the patients, the DSI and WHOQOL-Bref-TR scales will be filled in by the researcher. No procedure will be applied, they will receive routine hemodialysis treatment.
2. nd and 3rd Applications will be performed one week apart and the DSI and WHOQOL-Bref-TR will be filled in after the hemodialysis treatment without any procedure.

Statistics: SPSS Statistical Software program will be used for statistical analyses. While evaluating the study data, descriptive statistical methods (Mean, Standard deviation, median, frequency, ratio) as well as the Shapiro Wilk test and box plot graphics will be used for the normal distribution of the variables.

In the comparison of variables showing normal distribution between groups, ANOVA, Kruskal-Wallis H test, Tukey's post-hoc test, Pearson's chi-square test, Fisher's exact chi-square test, Bonferroni test, and multiple regression model analyses. Significance will be evaluated at p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Being diagnosed with ESRD,
* Being on hemodialysis for at least 3 months,
* Not having any sensory loss related to vision or hearing,
* Not having a psychiatric disease,
* Being open to communication and cooperation,
* Being willing to participate in the research

Exclusion Criteria:

* Being under 18 years of age,
* Not being in the end stage of chronic kidney disease,
* Receiving hemodialysis treatment for less than 3 months,
* Having sensory loss related to vision and hearing,
* Having a psychiatric disease,
* Not being open to communication and cooperation,
* Not volunteering to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
Dialysis Symptom Index (DSI) | This form was completed by each patient three times in total, at one-week intervals
  It was developed by Hemodialysis patients in order to determine the symptoms experienced by Hemodialysis patients and the level of impact on the patient. The scale, developed from the Memorial Symptom Diagnosis Scale Short Form, consists of 30 items. Responses are obtained on a 5-point Likert scale. The total scale score is obtained by adding up the scores obtained. This value varies between "0-15 0". The value "0" indicates that there is no symptom. The increase in the total points given to the answers towards 150 points shows that the effect of the mentioned symptom is increasing. The internal consistency coefficient of the scale was determined as 0.84.

SECONDARY OUTCOMES:
World Health Organization Quality of Life - Bref | This form was completed by each patient three times in total, at one-week intervals
  World Health Organization Quality of Life Bref is the short version of the WHOQOL-100 to assess the health-related quality of life, which has efficient psychometric properties, valid and reliable for Turkish society. It is essential for epidemiological survey and international report has built for psychometric properties for 26 country where Turkey within. It has 4 domains; physical health, psychology, social relations and environment. Each question is answered on a 5-point Likert scale. The raw score is converted into a percentage system. The quality of life is interpreted as good as it gets closer to 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Ecehan Bulut, Principal Investigator — PhD student
Locations (1):
- Kırklareli Eğitim ve Araştırma Hastanesi, Kırklareli, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No